CLINICAL TRIAL: NCT05889702
Title: Evaluation of the Kentucky Access to Recovery (KATR) Linkage Strategy
Brief Title: Kentucky Access to Recovery Evaluation
Status: Completed | Type: Observational
Sponsor: Terry Bunn (Other)
Responsible Party: Sponsor-Investigator, Terry Bunn, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 81811; R01CE003513-01-00 (Other Grant/Funding Number: CDC); R01CE003513-01 (NIH)
Record Dates: First submitted 2023-05-23; First posted 2023-06-05 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Substance Use Disorders; Treatment Adherence and Compliance
Keywords: Support Services; Recovery; Opioid Overdose; Addiction; Social Services; Appalachia
MeSH Terms: conditions — Substance-Related Disorders; Treatment Adherence and Compliance; Opiate Overdose; Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- KATR Clients: participants in the early stages of recovery and in substance use disorder (SUD) treatment; or those that have completed within the past year SUD treatment for opioid use disorder or stimulant use disorder or have a history of overdose from opioid use.
  Interventions: Behavioral: KATR Linkage Strategy

INTERVENTIONS:
Behavioral: KATR Linkage Strategy — The Kentucky ATR (KATR) strategy is a 25-county program that links county residents at or below the 200% national poverty level who have an illicit SUD and are in treatment or early recovery to evidence-based RSSs such as recovery housing, and to other RSSs.
  The KATR linkage approach uses vouchers as a linkage strategy for individuals in SUD treatment who have no other funding options to acquire critical RSSs. As such, KATR's linkage through vouchers is a "last resort" approach for linking to RSSs.

SUMMARY:
Evaluate the long-term effectiveness of implementing vouchers as a linkage strategy in a population requiring recovery support services (RSS) when no other funding sources are available. A within-subjects study design will be used to test the effectiveness of the Kentucky Access to Recovery (KATR) last resort voucher linkage approach to reduce the risk of nonfatal and fatal overdoses by (a) increasing an individual's recovery capital; (b) reducing resumption of illicit substance use; and (c) promoting relinking to RSSs if illicit substance use is resumed.

ELIGIBILITY:
Inclusion Criteria:

* be in SUD treatment or have completed within the past year SUD treatment for opioid use disorder or stimulant use disorder or have a history of overdose from opioid use
* be a first-time participant in KATR
* be in early stages of recovery (less than one year in recovery)
* be a resident of a KATR service county
* be at or below the 200% federal poverty level
* not have financial resources available through other funding mechanisms for RSSs
* be 18 years of age and older
* be in need of recovery supports that will enhance their likelihood of staying in recovery

Exclusion Criteria:

* Under 18
* Participated in KATR previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals in underserved areas with incomes at or below the 200% poverty level, individuals with prior criminal-justice involvement, veterans, and pregnant and parenting populations, with illicit SUD
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Change in Recovery Capital per person | Enrollment, Up to 6 months, 3 months post discharge, and 12 months post enrollment
  Recovery capital will be assessed using the Brief Assessment of Recovery Capital-10 (BARC-10); 10 item survey unidimensional measure of recovery capital, scores may range from 6-60 at any given time. Evaluation of the measure suggests that individuals who have a higher score are likely to reach or sustain a year or longer of recovery from substance use disorder.
Change in number of drug overdoses per person | Enrollment, Up to 6 months, 3 months post discharge, and 12 months post enrollment
  Number of drug overdoses will be assessed with the following survey question: In the past 30 days, did you experience an overdose or take too much of a substance that resulted in needing supervision or medical attention?
Change in number of days of illicit substance use per person | Enrollment, Up to 6 months, 3 months post discharge, and 12 months post enrollment
  Number of days illicit substance use will be assessed with the following survey question: During the past 30 days, how many days have you used any substance

CONTACTS AND LOCATIONS:
Overall Officials: Terry Bunn, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - FAHE, Berea, Kentucky
  - University of Kentucky, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No